CLINICAL TRIAL: NCT03067935
Title: Individual Patient Expanded Access-Glembatumumab Vedotin
Status: No longer available | Type: Expanded Access
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: Glembatumumab vedotin CU
Record Dates: First submitted 2017-02-23; First posted 2017-03-01 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Metastatic gpNMB Expressing Triple Negative Breast Cancer
MeSH Terms: interventions — glembatumumab vedotin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: glembatumumab vedotin

SUMMARY:
Celldex endeavors to make investigational products available to patients with life-threatening diseases who have exhausted other treatment options and where there is a reasonable expectation of benefit over risk. Requests for expanded access to glembatumumab vedotin in patients with gpNMB expressing triple negative breast cancer will be considered.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is 18 years of age or older.
2. The patient has histologically confirmed, gpNMB expressing, metastatic triple-negative breast cancer
3. Overexpression of gpNMB in at least one tumor sample as determined by a Sponsor approved laboratory using IHC methods
4. The patient does not have abnormal organ function, active autoimmune disease, active infections or additional concurrent conditions that would compromise the patient's ability to safely receive glembatumumb vedotin.
5. The patient is not eligible for or cannot access ongoing glembatumumab vedotin clinical trials
6. The patient does not qualify for, or cannot access, other comparable or satisfactory alternative therapy for triple negative breast cancer.
7. The patient is able to read and understand, and has signed a patient informed consent form, which outlines the nature of the proposed treatment and the anticipated benefits and risks of treatment with glembatumumab vedotin.

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar composition to glembatumumab vedotin, MMAE, dolastatin or auristatin.
2. Pregnant or breast-feeding women, and women or men who are not willing to use effective contraception during the time from signing of informed consent through two months after the last dose of glembatumumab vedotin treatment.
3. The patient was previously treated with glembatumumab vedotin or previously enrolled on the METRIC trial (regardless of which arm they were randomized to).
4. Any underlying medical condition that, in the investigator's or Sponsor's opinion, will make the administration of Glembatumumab vedotin hazardous to the patient, or would obscure the interpretation of adverse events.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult